CLINICAL TRIAL: NCT07231432
Title: Promoting Community-based Kangaroo Care Among Mothers of Low Birth Weight Infants in Rural India
Brief Title: Promoting Kangaroo Care for Preterm or Low Birthweight Infants in Rural India
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nisha Fahey, Assistant Professor of Pediatrics, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: K23HD112602 (NIH); K23HD112602-01A1 (NIH)
Record Dates: First submitted 2025-11-12; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Preterm Birth; Skin to Skin Contact; Low Birth Weight; Kangaroo Care
MeSH Terms: conditions — Premature Birth | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Aim 1 consists of focus groups and qualitative analysis. Aim 2 consists of pilot testing interventions. Aim 3 includes the interventional study model, which is described here. As a part of the Multiphase Optimization Strategy (MOST) design-based trial, Aim 3 consists of an optimization trial using full factorial design to test combinations of intervention components, known as experimental conditions, and identify key combinations to include in an optimized, multicomponent intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Base Intervention + Behavioral Interventions A + B + C (Experimental)
  Interventions: Behavioral: Behavioral Interventions
- Base Intervention + Behavioral Interventions A + B (Experimental)
  Interventions: Behavioral: Behavioral Interventions
- Base Intervention + Behavioral Interventions A + C (Experimental)
  Interventions: Behavioral: Behavioral Interventions
- Base Intervention + Behavioral Intervention A (Experimental)
  Interventions: Behavioral: Behavioral Interventions
- Base Intervention + Behavioral Interventions B + C (Experimental)
  Interventions: Behavioral: Behavioral Interventions
- Base Intervention + Behavioral Intervention B (Experimental)
  Interventions: Behavioral: Behavioral Interventions
- Base Intervention + Behavioral Intervention C (Experimental)
  Interventions: Behavioral: Behavioral Interventions
- Base Intervention + No Experimental Behavioral Interventions (No Intervention)

INTERVENTIONS:
Behavioral: Behavioral Interventions — The interventions have not been determined yet. The intervention aspect of the study is not active at this time. This information will be updated at a later time to include more details.
  Arms: Base Intervention + Behavioral Intervention A; Base Intervention + Behavioral Intervention B; Base Intervention + Behavioral Intervention C; Base Intervention + Behavioral Interventions A + B; Base Intervention + Behavioral Interventions A + B + C; Base Intervention + Behavioral Interventions A + C; Base Intervention + Behavioral Interventions B + C

SUMMARY:
The goal of this study is to develop ways to help mothers of preterm or low birth weight infants do Kangaroo Care at home after discharge from the Neonatal Intensive Care Unit in rural India.

DETAILED DESCRIPTION:
This study aims to create and evaluate interventions to support the practice of Kangaroo Care among mothers of preterm or low birth weight infants in the community-seeing after discharge from the Neonatal Intensive Care Unity. Using a mixed methods and Multiphase Optimization Strategy (MOST) design-based trial, we aim to: Aim 1: Use community-engaged research and qualitative methods to refine up to four individual candidate interventions to overcome barriers to community-based Kangaroo Care, Aim 2: Pilot individual candidate interventions to assess implementation outcomes and define optimization criterion tailored for the community setting, Aim 3: Conduct a MOST design-based optimization trial to develop a community-informed, multicomponent intervention to promote community-based Kangaroo Care

ELIGIBILITY:
AIM 1

Mothers

* Mothers of former low birthweight (<2500 grams at birth) infants who were hospitalized in the Shree Krishna Hospital NICU
* Performed Kangaroo Care during their infant's hospitalization
* Live in a village that is "adopted" by and within a 50-kilometer radius of Shree Krishna Hospital
* At least 18 years old
* Speak Gujarati

Healthcare Providers- Physicians:

* Physicians and nurses who work in either the Shree Krishna Hospital NICU or in community settings within a 50-kilometer radius who provide newborn care to at least 3 newborns each week
* At least 18 years old
* Speak Gujarati

Village Health Workers:

* Village health workers who operate in one of the "adopted" villages within a 50-kilometer radius of Shree Krishna Hospital
* We will aim to recruit one health worker from 10 of the 15 subregions of the district of Anand, based on geography
* At least 18 years old
* Speak Gujarati

AIM 2

Mothers:

* Mothers of an infant born with low birthweight (< 2500g) who is hospitalized in the NICU at Shree Krishna Hospital with an anticipated discharge weight of less than 2500g
* Must reside in a village "adopted" by and within a 50-kilometer radius of Shree Krishna Hospital and plan to live there for at least 6 weeks after NICU discharge
* Speaks Gujarati
* At least 18 years old

AIM 3

Mothers:

* Mothers of an infant born with low birthweight (< 2500g) who is hospitalized in the NICU at Shree Krishna Hospital with an anticipated discharge weight of less than 2500g
* Must reside in a village "adopted" by and within a 50-kilometer radius of Shree Krishna Hospital and plan to live there for at least 6 weeks after NICU discharge
* Speaks Gujarati
* At least 18 years old

Exclusion Criteria (applicable to all aims)

* Persons unable to provide informed consent
* Pregnant women may enroll in this study, though, we will not be intentionally recruiting pregnant women. (Refer to section 18 for more information on this)
* Prisoners will not be included in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2028-08-13 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Uptake of community-based Kangaroo Care use | 6 weeks
  Self-report of any Kangaroo Care at home after NICU discharge

SECONDARY OUTCOMES:
Maternal Intention to perform Kangaroo Care | Baseline (day 0)
  Self-report of intention to perform Kangaroo Care at home
Maternal Self-Efficacy to perform Kangaroo Care | 6 weeks
  Maternal Self-Efficacy Scale questionnaire
Adherence to community-based Kangaroo Care | 6 weeks
  Self-report of the last date Kangaroo Care was performed at home
Frequency of community-based Kangaroo Care use | 6 weeks
  Self-report of number of days Kangaroo Care was provided at home
Acceptability of the intervention | 6 weeks
  Client Satisfaction Questionnaire
Appropriateness of the intervention | 6 weeks
  Qualitative Exit Interview with a trained member of the research staff
Material Costs of the intervention | 6 weeks
  Cumulative cost of intervention delivery per participant
Engagement with the intervention | 6 weeks
  Self-reported engagement with intervention (# of instances)
Feasibility of the intervention | 6 weeks
  Feasibility of Intervention Measure questionnaire
Usability of the intervention | 6 weeks
  System Usability Scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nisha Fahey, DO, MSc, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Sufficient data from this project will be preserved to validate and replicate research findings described in the Aims. The final dataset will include self-reported demographics, behavioral beliefs, acceptability, appropriateness, material costs, engagement, feasibility, usability, uptake, frequency, and adherence. Additional data sets will include coded qualitative data. We will share de-identified individual participant-level data.
Supporting Information: Study Protocol
Time Frame: All scientific data that can be shared from this project will be made available as soon as possible, and no later than 12 months of the end of the funding period. The duration of preservation and sharing of the data will be a minimum of 10 years after the funding period.
Access Criteria: All dataset(s) that can be shared, along with related metadata, will be deposited in the Harvard Dataverse Repository (https://dataverse.harvard.edu/). This will ensure the research community has long-term access to the data. Dataverse provides a DOI for the dataset related to this project, providing permanent identification for the data and ensuring that it will always be found with the same DOI. Its software platform provides a preservation and archival infrastructure and allows researchers to share, keep control of, and get recognition for their data through an easy-to-access web browser interface.